CLINICAL TRIAL: NCT06044155
Title: Efficacy and Safety After Failure of a First POEM
Brief Title: redoPOEM : Failure of a First POEM
Acronym: redoPOEM
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/17
Record Dates: First submitted 2023-08-10; First posted 2023-09-21 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Achalasia
Keywords: achalasia; redoPOEM; POEM; per-oral endoscopic myotomy; retrospective; multicenter; efficacy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
observational study, measurement of efficacy in the cohort.

DETAILED DESCRIPTION:
Achalasia is a motor disorder of the esophagus with a prevalence of 1/10000. Multiple treatments have been proposed, including endoscopic dilation, botulinum toxin injection and surgery using the Heller myotomy technique. These techniques are moderately effective and/or carry the risk of per- and post-procedural complications. POEM has been available since 2008, with 80-90% efficacy and 90% safety, and no serious complications have been reported. In the event of failure of a first POEM, a second POEM, known as "redoPOEM", can be proposed. Several studies show efficacy of between 76% and 96% and a safety of between 80% and 86%, with only one serious adverse event reported, and no deaths. However, the studies carried out involved small numbers of patients, generally around 50, the vast majority in Asian countries. The aim of this study was therefore to evaluate the efficacy and safety of redoPOEM reported in patients from several expert centers in Europe.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* diagnosis of achalasia based on clinical criteria according to Eckardt score, manometry, and radiology when available.
* failure after POEM (Eckardt score > or equal to 4 in consultation) treated with a new POEM.
* no active digestive neoplasia.

Exclusion Criteria:

* Technical failure of redoPOEM
* Person not affiliated to a Social Security scheme
* Language barrier preventing fair collection of non-opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with achalasia and failure after POEM treated with a new POEM
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Efficacy : score of Eckardt | 3 months after redoPOEM
  Evaluation of Eckardt score at 3 months after redoPOEM strictly less than 4. Each question is rated from 0 to 3. It consists of 4 items with a total score varies from 0 to 12.

SECONDARY OUTCOMES:
Safety : Number of adverse events of grade II | Through study completion, an average of 1 year
  Evaluation of absence of adverse events of grade II or higher according to AGREE classification.
Efficacy : Number of Eckart score strictly below 4 | Through study completion, an average of 1 year
  Evaluation of Eckardt score strictly below 4 at last known follow-up after redoPOEM. Each question is rated from 0 to 3. It consists of 4 items with a total score varies from 0 to 12.
Efficacy : Number of new additional procedure | Through study completion, an average of 1 year
  Evaluation of number of an additional procedure because of failure of redoPOEM.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur BERGER, MD, Principal Investigator — University Hospital, Bordeaux
Locations (14):
- France (14):
  - Chu de Bordeaux, Bordeaux
  - Clinique des Cèdres, Cornebarrieu
  - CHU Dijon Bourgogne, Dijon
  - Centre Hospitalier Intercommunal de Toulon - La Seyne-sur-Mer, La Seyne-sur-Mer
  - CHU Lille, Lille
  - CHU de Limoges, Limoges
  - Hospices civils de Lyon, Lyon
  - Hôpitaux Universitaires de Marseille Nord, Marseille
  - CHU de Nantes, Nantes
  - CHU de Nice - Hôpital Archet, Nice
  - CHU de Nîmes, Nîmes
  - AP-HP Hôpital Cochin, Paris
  - CHU de Rennes, Rennes
  - CHRU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Angelo A, Pioche M, Barret M, Gonzalez JM, Wallenhorst T, Coron E, Velut G, Vanbiervliet G, Onana Ndong P, Jacques J, Schaefer M, Levy J, Caillo L, Rahmi G, Aidibi A, Ah-Soune P, Degand T, Saunier M, Zerbib F, Berger A. RedoPOEM: efficacy and safety after failure of a first POEM for esophageal motility disorders. Surg Endosc. 2026 Jan 23. doi: 10.1007/s00464-026-12564-4. Online ahead of print. PMID 41575544